CLINICAL TRIAL: NCT04492241
Title: Evaluation of Efficacy and Safety of Ginkgo Leaf Extract and Armillariella Mellea Powder Oral Solution for the Treatment of Motoric Cognitive Risk Syndrome: A Multi-centre, Randomised, Double Blind and Placebo-controlled Study
Brief Title: Ginkgo Leaf Extract and Armillariella Mellea Powder Oral Solution for the Treatment of Motoric Cognitive Risk Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Beijing Stroke Association (Unknown)
Responsible Party: Principal Investigator, Jingjing Li, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY2020-052-03
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Motoric Cognitive Risk Syndrome; Mild Cognitive Impairment; Aging; Locomotive Syndrome
Keywords: MCR; Ginkgo Leaf Extract; Armillariella Mellea Powder; MCI
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Ginkgo biloba extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Arm (Experimental): Ginkgo Leaf Extract and Armillariella Mellea Powder Oral Solution, TID
  Interventions: Drug: Ginkgo Leaf Extract and Armillariella Mellea Powder Oral Solution
- Control Arm (Placebo Comparator): Simulation of Ginkgo Leaf Extract and Armillariella Mellea Powder Oral Solution, TID
  Interventions: Drug: Simulation of Ginkgo Leaf Extract and Armillariella Mellea Powder Oral Solution

INTERVENTIONS:
Drug: Ginkgo Leaf Extract and Armillariella Mellea Powder Oral Solution — TID for 6 month after enrolment Glass oral bottle, 10 ml/bottle. Study Arm Component: Ginkgo Leaf Extract and Armillariella Mellea Powder, konjac (sweetener), purified water.
  Other Names: Yinxingmihuan Koufuyongye
  Arms: Study Arm
Drug: Simulation of Ginkgo Leaf Extract and Armillariella Mellea Powder Oral Solution — TID for 6 month after enrolment Glass oral bottle, 10 ml/bottle. Placebo Arm Component: Caramel color (food color), konjac (sweetener), sucrose octaacetate (food additive), sodium benzoate (food additive), purified water.
  Other Names: Yinxingmihuan Koufuyongye Moniji
  Arms: Control Arm

SUMMARY:
This is a multi-centre, randomised, double blind, placebo controlled study on participants with Motoric Cognitive Risk Syndrome to evaluate the efficacy and safety of Ginkgo Leaf Extract and Armillariella Mellea Powder Oral Solution.

DETAILED DESCRIPTION:
Cognition and locomotion are two human abilities controlled by the brain. Their decline is highly prevalent with aging, and is greater than the simple sum of their respective prevalence, suggesting a complex age-related interplay between cognition and locomotion.

Recently, a systematic review and meta-analysis has provided evidence that poor gait performance predicts dementia and, in particular, has demonstrated that "motoric cognitive risk" (MCR) syndrome, which has been described in cognitively healthy individuals and combines subjective cognitive complaint with objective slow gait speed, is a pre-dementia syndrome.

MCR as a relatively new recognised clinical syndrome is with a high prevalence calculated around 10% in world population aged 60 and above. MCR syndrome predicts mild and major neurocognitive disorders. MCR syndrome does not rely on a complex and time-consuming assessment, making it applicable to the aging population. Thus, MCR syndrome seems to be a good syndrome to identify individuals at risk of mild and major neurocognitive disorders in any type of healthcare setting.

Ginkgo Leaf Extract and Armillariella Mellea Powder Oral Solution has proven efficacy for cognitive function deterioration in preliminary studies. The aim of this study is to evaluate its efficacy and safety for MCR.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form
* Capability of independent living (capability of dressing, bathing, walking, and bed-chair transfer)
* Met Motoric Cognitive Risk Syndrome (MCR) criteria:

Single task slow gait ( male 60 to 74 y, gait <75.4 cm/s; male ≥ 75 y, gait < 59.1 cm/s; female 60 to 74 y, gait <70.0 cm/s; female ≥ 75 y, gait < 48.3 cm/s) And The Montreal Cognitive Assessment (MoCA) ≤ 26 (≥ 12 education year) or MoCA ≤ 25 (< 12 education year)

* Anticipated good compliance per protocol

Exclusion Criteria:

* Illiteracy
* The Mini-Mental State Examination (MMSE) ≤ 23
* Medical history of mental illness such as schizophrenia, severe anxiety and depression.
* Medical history of Alzheimer's disease, Parkinson's disease, frontotemporal dementia or Huntington's disease.
* Dementia caused by other causes (such as central nervous system trauma, tumor, infection, metabolic disease, normal pressure hydrocephalus, folic acid, vitamin B12 deficiency, thyroid Inferior functions, etc.).
* History of epilepsy, or taking anti-epileptic drugs.
* History of myocardial infarction or stroke
* History of malignant tumor
* Coagulation disorder, systemic bleeding; or previous coagulation disorder or systemic bleeding disease history.
* History of thrombocytopenia or neutropenia.
* History of blood system diseases or liver function abnormalities caused by medication
* Contraindications to ginkgo drugs and a history of known allergies.
* Aphasia, severe hearing or visual impairment, dominant hemiplegia, and other impacts on cognitive evaluation The status of the test.
* Known slow gait causes (non-neurological causes [such as: arthritis, heart disease] and neurological causes [bias Paralysis, ataxia, spasticity, Parkinson's disease and frontal lobe disease])
* Severe heart and lung diseases (coronary heart disease, LVEF<40%, NYHA heart failure grade ≥III, asthma asthma).
* Severe arrhythmia, heart rate >120bpm or <50bpm. (17) Blood pressure <90/60mmHg
* Severe anemia, Hb<100g/L
* Severe liver or renal insufficiency (ALT > 2 times the upper limit of normal or AST > 2 times the upper limit of normal; Creatinine >1.5 times the upper limit of normal)
* Leukopenia (<2×109/l) or thrombocytopenia (<100×109/l)
* Currently enrolled in other drug or medical device study
* Planned any surgery within 6 months at screening
* Considered by investigators as unsuitable participant of this study

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2021-07-05 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of ADAS-Cog | 6 month after enrolment
  The Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) test is one of the most frequently used tests to measure cognition in research studies and clinical trials for new drugs and other interventions.The test administrator adds up points for the errors in each task of the ADAS-Cog for a total score ranging from 0 to 70. The greater the dysfunction, the greater the score. A score of 70 represents the most severe impairment and 0 represents the least impairment.

SECONDARY OUTCOMES:
Frequency of Falls | 6 month after enrolment
  Fall refers to sudden, involuntary, unintentional body position change, falling to the ground or lower plane. Falls include the following two types: (1) falls from one plane to another; (2) falls on the same plane.
Change of each items from ADAS-Cog | 6 month after enrolment
  The Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog): A score of 70 represents the most severe impairment and 0 represents the least impairment. The 12 items of ADAS-Cog applied in this study: Word Recall, Commands, Constructional Praxis, Naming, Ideational Praxis, Orientation, Word Recognition, Remembering Word Recognition Test Instructions, Comprehension of Spoken Language, Word-Finding Difficulty, Spoken Language Ability, Concentration/Distractibility
Percentage of change of ADAS-Cog score 4 or more | 6 month after enrolment
  The Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog): A score of 70 represents the most severe impairment and 0 represents the least impairment. Comparing to baseline, the percentage of ADAS-Cog score decreased 4 or more
TMT-A Score | 6 month after enrolment
  Trail Making Test (TMT) Parts A & B. Both parts of the Trail Making Test consist of 25 circles distributed over a sheet of paper. In Part A, the circles are numbered 1 - 25, and the patient should draw lines to connect the numbers in ascending order.
TMT-B Score | 6 month after enrolment
  Trail Making Test (TMT) Parts A & B. Both parts of the Trail Making Test consist of 25 circles distributed over a sheet of paper. In Part B, the circles include both numbers (1 - 13) and letters (A - L); as in Part A, the patient draws lines to connect the circles in an ascending pattern, but with the added task of alternating between the numbers and letters (i.e., 1-A-2-B-3-C, etc.).
Functional Activities Questionnaire score | 6 month after enrolment
  Sum scores (range 0-30). Cutpoint of 9 (dependent in 3 or more activities) is recommended to indicate impaired function and possible cognitive impairment.
Activities of Daily Living (ADLs) score | 6 month after enrolment
  ADL self-performance measures what the resident actually did (not what he or she might be capable of doing) within each ADL category over the prior seven days, according to a performance-based scale. ADL self-performance coding ranges from 0 (independent) to 4 (total dependence) and is coded as 20 items. The total ADL score is a very important component of the RUG categories and is calculated from the seven days immediately preceding and including the date of the assessment. Chang- es, including improvements and declines in function that have occurred since the assessment date are not considered when coding the MDS.
The Neuropsychiatric Inventory Questionnaire | 6 month after enrolment
  The Neuropsychiatric Inventory-Questionnaire (NPI-Q) was developed and cross- validated with the standard NPI to provide a brief assessment of neuropsychiatric symptomatology in routine clinical practice settings. The NPI-Q is designed to be a self-administered questionnaire completed by informants about patients for whom they care. Each of the 12 NPI-Q domains contains a survey question that reflects cardinal symptoms of that domain.
Dementia Conversion Rate | 6 month after enrolment
  Defined as conversion rate of MMSE≤23 at 6 month. The Mini-Mental State Examination (MMSE) is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. It is commonly used in medicine and allied health to screen for dementia.
  It is also used to estimate the severity and progression of cognitive impairment and to follow the course of cognitive changes in an individual over time; thus making it an effective way to document an individual's response to treatment. The MMSE's purpose has been not, on its own, to provide a diagnosis for any particular nosological entity.
Single-task gait speed test | 6 month after enrolment
  The test can be performed with any patient able to walk 4 metres using the instructions below:
  1. Instruct the patient to walk at their normal pace. Patients may use an assistive device, if needed.
  2. Ask the patient to walk down a hallway through a 1-metre zone for acceleration, a central 4- metre "testing" zone, and a 1-metre zone for deceleration (the patient should not start to slow down before the 4-metre mark).
  3. Start the timer with the first footfall after the 0-metre line.
  4. Stop the timer with the first footfall after the 4-metre line.
Dual-task gait speed test-naming animals | 6 month after enrolment
  For the dual-task trials, participants walked the length of 4 metres while subtracting serial 7s from 100 aloud or while naming animals aloud.

OTHER OUTCOMES:
Safety endpoints: major cerebral-cardiovascular events | 6 month after enrolment
  Defined as any non-fatal acute myocardial infarction, non-fatal stroke, cardiovascular death.
Adverse Drug Reaction | 6 month after enrolment
  An adverse drug reaction is a harmful reaction to a medicine given at the correct dose.

CONTACTS AND LOCATIONS:
Overall Officials: Xingquan Zhao, PhD, Study Chair — Department of Neurology, Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China